CLINICAL TRIAL: NCT01215201
Title: Adjunctive Non-Surgical Therapy of Inflamed Periodontal Pockets Using Diode Lasers During Maintenance Therapy
Brief Title: Diode Laser Study for Periodontal Maintenance Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0452-09-EP
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Periodontal Diseases; Periodontitis, Apical, Chronic Nonsuppurative; Suppuration of Gingival Crevice
Keywords: Periodontal maintenance; ≥5mm probing depth; bleeding on probing and/or suppuration
MeSH Terms: conditions — Periodontal Diseases; Periapical Granuloma | interventions — Tooth Exfoliation; Root Planing; Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scaling and Root Planing Alone (Other): Control group
  Interventions: Procedure: Scaling and Root Planing
- Diode Laser plus Scaling and Root Planing (Experimental): Diode Laser is used in addition to Scaling and root planing procedure.
  Interventions: Procedure: Diode Laser + Scaling and Root Planing

INTERVENTIONS:
Procedure: Scaling and Root Planing — Use periodontal hand instruments (curettes) to remove plaque, bacteria, and deposits on the root's surfaces.
  Arms: Scaling and Root Planing Alone
Procedure: Diode Laser + Scaling and Root Planing — First: Periodontal hand instruments (curettes) were used to remove plaque, bacteria, and deposits on the root's surfaces (within a periodontal pocket) Then: Biolase 940 nm Ezlase diode laser was used to sterilize a periodontal pocket. Power: 0.80 Watts Wavelength: 940 nm Energy level: 0.80 Joules/second Mode of beam delivery: continuous
  Arms: Diode Laser plus Scaling and Root Planing

SUMMARY:
This study tries to determine whether the additional use of laser with "cleaning" (known as scaling and root planning) will result in the reduction of inflammation, reduction of bleeding upon examination and reduction of pocket depth in patients who are being maintained on a regular basis but have pocket depths that are ≥5mm with bleeding. When a pocket is bleeding, it is inflamed. It is usually "cleaned" with periodontal instruments (root-planed) to establish health. Some research also advocates using laser therapy to treat a bleeding pocket. Laser therapy is presently being performed in some dental offices and dental colleges. This research is trying to see if the additional laser therapy is beneficial.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the adjunctive use of diode laser with scaling and root planing is more effective than scaling and root planing alone in clinically reducing periodontal pocket depth (PD), reducing bleeding on probing (BOP) and gaining of clinical attachment level (CAL). It also assesses whether diode laser with scaling and root planing will have an effect on cytokines and inflammatory biomarkers compared to root planing alone.

Any adult who is currently a routine periodontal maintenance patient and has one or more ≥ 5mm pockets with BOP will be invited to participate in the study. If they choose to participate, they will sign an informed consent. Crevicular fluid samples from each test site and another non-involved site in the mouth will be collected utilizing the standard protocol and frozen for later analyses of the presence of certain inflammatory biomarkers (IL-1β). Baseline data (i.e., PD, CAL, BOP, suppuration, supragingival plaque, subgingival restorative margins, smoking status) will be collected. The involved teeth will then be randomly treated with scaling and root-planing with hand instruments and diode laser (test) or scaling and root-planing with hand instruments alone. The patient will return 3 months later for follow-up data collection. He/she will then receive his/her regular 3 month maintenance therapy.

The changes between baseline and 3 months for the clinical parameters and gingival crevicular fluids' inflammatory biomarkers will be compared between test and control experimental sites.

ELIGIBILITY:
Inclusion Criteria:

* Any adult periodontal maintenance patient having had chronic periodontitis with last active therapy at least 3 months prior and with 1 or more sites/subject with ≥5mm probing depth that have bleeding on probing and/or suppuration. They have signed an informed consent form to participate in the study.

Exclusion Criteria:

* Subjects who are un-controlled diabetics, use NSAIDS regularly for chronic disease/pain, used antibiotics for the last 3 months, require antibiotic coverage for therapy, are pregnant and below age 30.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2011-06-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
Periodontal clinical parameters | 3 months
  Reduction in Probing Depth, Gaining of clinical attachment level, Reduction of Bleeding upon Probing, Reduction of Plaque accumulation, reduction of IL-1B inflammatory marker.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi-Trang Nguyen, DDS, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Dentistry, Lincoln, Nebraska, United States